CLINICAL TRIAL: NCT00562692
Title: Role of Natriuretic Peptides in the Treatment of Acutely Decompensated Heart Failure Patient With Obstructive Airways Disease
Acronym: BNP in OAD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment very difficult. Study drug expired so we have stopped the study.
Sponsor: The Alfred (Other)
Collaborators: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Principal Investigator, Henry Krum, Head Clinical Pharmacology, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-02/05; Project No. 11/06
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure
Keywords: Heart failure; OAD; BNP; Heart Failure patients who present to the emergency department
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Nesiritide
  Interventions: Drug: Nesiritide
- B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nesiritide — Nesiritide 4 hour infusion
  Arms: A
Drug: Placebo — Placebo infusion
  Arms: B

SUMMARY:
Brain natriuretic peptide (BNP) is a useful therapy when treating patients with heart failure. As many of these patients also have airways disease it is important to determine if BNP also has a positive effect on their respiratory condition. The role of BNP in airways disease has never been studied although there is evidence to suggest that it will have a positive effect.

The current study is therefore a proof on concept study which will demonstrate whether BNP (nesiritide) will improve both heart failure and airflow obstruction in patient who have both.

The investigators are looking to enroll 40 patients with heart failure and airways disease who present to hospital emergency departments. Patients who consent and meet the entry criteria will be randomised to receive either nesiritide or placebo in addition to standard therapy. They will receive a bolus of study medication followed by a 4 hour infusion. Before, at hourly intervals and immediately following the infusion the following data will be collected:

* dyspnoea score
* respiratory rate
* FEV1 (if able to be performed)
* peak respiratory flow rates (PEFR, if able to be performed)
* requirement for concomitant bronchodilator therapy
* urinary GMP At all times during the study period and at the conclusion of the study patients will be provided with the best available therapy for their condition at the physicians' discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Over 18 years of age
3. Confirmed written informed consent.
4. Acute decompensated heart failure based on physicians assessment and requiring treatment as per standard emergency department protocols for this condition.
5. Requirement for intravenous therapy of HF, e.g. diuretic, vasodilator.
6. COAD based on physician's assessment and requiring treatment as per standard emergency department protocols for this condition. Must have at least 2 of the following criteria:

   * history of smoking > 20 pack years,
   * prior history of PFTs within last 1 year consistent with COAD,
   * history of chronic cough and sputum production,
   * progressive dyspnea, episodes of acute bronchitis over at least 2 yrs

Exclusion Criteria:

1. Women lactating, pregnant or of childbearing potential not using 2 reliable contraceptive methods.
2. Patients who had received an investigational new drug within the last 4 weeks.
3. Patients with a history of a psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study.
4. SBP <90mmHg
5. Creatinine >0.25mmol/L
6. Sp02 < 80% on supplemental oxygen or known cor pulmonale with TR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To compare the need for and the length of time patients require non invasive ventilation when treated with nesiritide vs placebo. | 24 hours

SECONDARY OUTCOMES:
dyspnoea score respiratory rate FEV1 PEFR requirement for concomitant bronchodilator therapy BNP | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS FRACP PhD, Principal Investigator — Monash University / Alfred Hospital; Peter Cameron, Principal Investigator — Monash University / Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia